CLINICAL TRIAL: NCT04120051
Title: The SIMBA Project - The Effect of a Prebiotic Supplement on Glucose Metabolism and Gut Microbiota
Brief Title: The SIMBA Project - The Effect of a Prebiotic Supplement on Glucose Metabolism and Gut Microbiota in Obese Adults
Acronym: SIMBA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: FermBiotics ApS (Unknown)
Responsible Party: Principal Investigator, Mads Vendelbo Lind, Post doc, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: H-19041432
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Glucose Metabolism; Metabolic Syndrome; Gut Microbiota
Keywords: Gut Microbiota; Metabolic syndrome; Obesity; Supplement
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to the Fermented Canola-Seaweed supplement or control and are expected to consume one sachet (5 grams) of either every day for 6 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization sequence will be done by an investigator without contact to the participants. The personnel conducting the study will allocate participants to the sequence of intervention using a list of participant identification numbers matched with allocated sequences. The participants will be blinded to the intervention and blinding of the allocation sequence will be present for investigators during sample analysis and initial data analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented canola-seaweed supplement (Experimental): Ingredients: Canola meal, seaweed, wheat, glucose, Vitamin D and lactic acid bacteria
  Interventions: Dietary Supplement: Fermented canola-seaweed
- Placebo (Placebo Comparator): Ingredients: Rye flour, water, iodized salt, brown sugar
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented canola-seaweed — A daily sachet with 5 gram FCS-granulate for 6 weeks
  Arms: Fermented canola-seaweed supplement
Other: Placebo — A daily sachet with 5 gram rye cereal for 6 weeks
  Arms: Placebo

SUMMARY:
Modulation of the gut microbiota via administration of pro- and prebiotics have been proposed to contribute to weight loss and reduce plasma glucose and serum lipid levels, improving the inflammatory state and decreasing the incidence of type 2 diabetes and cardiovascular disease. This study will test a fermented canola-seaweed (FCS) product, high in glucosinolates and putatively prebiotic oligosaccharides, in human subjects with obesity.

DETAILED DESCRIPTION:
The overall objective of this study is to investigate a fermented canola-seaweed (FCS) product in obese human subjects with increased risk of metabolic syndrome (MS). We will study the effects of the FCS on glucose handling and related cardiometabolic traits such as dyslipidemia and low-grade systemic inflammation. Finally, we will examine the gut microbiota and the metabolic phenotype of the subjects to explore molecular mechanisms related to the potential improvements.

It is hypothesized that the FCS product will improve postprandial glucose handling, blood lipids and low-grade inflammation in obese subjects with increased risk of MS. Furthermore, it is hypothesized that this effect is modified through gut microbiota compositional and functionality changes

Methods:

This study will be conducted as a randomized, controlled, investigator and participant blinded intervention trial. The participants will be randomized to the FCS supplement or control and are expected to consume one sachet of either every day for 6 weeks.

Randomization, blinding and allocation concealment:

After having given oral and written consent, randomization will be performed separately for each participant in blocks of variable size to ensure equal randomization throughout the enrolment phase of the study. The randomization sequence will be done by an investigator without contact to the participants. The personnel conducting the study will allocate participants to the sequence of intervention using a list of participant identification numbers matched with allocated sequences. The participants will be blinded to the intervention and blinding of the allocation sequence will be present for investigators during sample analysis and initial data analysis.

Examinations:

Participants will arrive for clinical examination after an overnight fast of at least 8 hours. Lifestyle questionnaires and questionnaires about medication use will be performed for baseline characterization of the participants. Blood pressure and anthropometric measurements are performed including measurements of body weight, height, waist and hip circumference, and bio-impedance measurements for assessing body fat mass. A fasting blood sample is obtained and an oral glucose tolerance test (OGTT) is performed with collection of blood samples after 0, 30 and 120 min. Samples will be analyzed with standard clinical procedures for glycaemic variability markers, including glucose, insulin, c-peptide, and HbA1c, as well as plasma lipids. Furthermore, fecal samples will be collected at both examination visits and kept stored for future microbiota analyses, using untargeted shotgun sequencing.

Samples in biobank will be stored for further analyses, which could include gastrointestinal hormones, gut microbiota metabolites, blood, and fecal metabolome and low-grade inflammation markers. In addition, a subgroup of participants (10 in each group) will be equipped with a 24-h continuous glucose monitoring device for 14 days at the start of the intervention period. Both examination days consists of similar examinations and data collections and are estimated to last approximately 2½ hours.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Age between 30 and 65 years
* Body mass index ≥31 kg/m^2

Exclusion Criteria:

* Body mass index <31 kg/m^2
* Diagnosis of diabetes (HbA1c ≥ 6,5% (48 mmol/mol)) or pharmacological treatment of diabetes
* Use of peroral glucocorticoids
* Lack of compliance with the procedures (ingestion of sachets) in the study protocol, judged by Investigator
* Ingestion of pre- or probiotic supplements during the study and 14 days prior to study start
* Use of systemic antibiotics 1 month prior to study start
* Use of cholesterol lowering drugs
* Have had an obesity or abdominal surgery
* Chronic inflammation disorders (excluding obesity)
* Diagnosed psychiatric disorder including depression requiring treatment
* Gastro intestinal and liver disorders
* Gluten intolerance
* Maltodextrin intolerance
* Intensive physical training/ elite athlete (>10 hours of strenuous physical activity per week)
* Pregnant or lactating
* High intake of alcohol (>14 drinks/week for women and >21 drinks/week for men)
* Simultaneous blood donation for other purpose than this study
* Simultaneous participation in other clinical intervention studies
* Inability, physically or mentally, to comply with the procedures required by the study protocol as evaluated by the principal investigator or clinical responsible.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
changes in 2-h post-OGTT glucose in blood between baseline and endpoint | Week 0 and Week 6
  2 hour post oral glucose tolerance test glucose measurement in blood (mmol/L)

SECONDARY OUTCOMES:
Changes in Hba1c between baseline and endpoint | Week 0 and Week 6
  fasting measurement of blood glycated hemoglobin (%)
Changes in fasting blood glucose between baseline and endpoint | Week 0 and Week 6
  Fasting measurement of blood glucose (mmol/L)
Changes in 30 min post OGTT between baseline and endpoint | Week 0 and Week 6
  Measurement of blood glucose 30 min after OGTT (mmol/L)
Insulin sensitivity and secretion | Week 0 and Week 6
  Measured as part of the OGTT. Plasma glucose (mmol/l). Plasma insulin - fasting (pmol/l)
Changes in blood lipids between baseline and endpoint | Week 0 and Week 6
  Measurements of total and HDL cholesterol (mmol/L) and triglycerides (mmol/L)
Changes in C-Reactive Protein between baseline and endpoint | Week 0 and Week 6
  Blood measurements of C-Reactive Protein (mg/L)
Changes in Interleukin-6 between baseline and endpoint | Week 0 and Week 6
  Blood measurements of Interleukin-6 (pg/mL)
Changes in small metabolites between baseline and endpoint | Week 0 and Week 6
  Measured using blood metabolomic measurements of amino acids, lipids, and other small metabolites (umol/L)
Changes in weight between baseline and endpoint | Week 0 and Week 6
  Measured using a Tanita body composition analyser. Body weight in kilograms
Changes in waist circumference between baseline and endpoint | Week 0 and Week 6
  Measured using measurement tape
Changes in body composition between baseline and endpoint | Week 0 and Week 6
  Measured using a Tanita body composition analyser. Fat free mass and Body fat mass in kilograms used to calculate body fat percentage.
Changes in blood pressure (BP) between baseline and endpoint | Week 0 and Week 6
  Systolic BP (mmHG) Diastolic BP (mmHG)
Continuous glucose monitoring | Week 0
  Continuous glucose monitor from Abbott is worn for 14 days in each period providing glucose measurements continuously (mmol/L)
Changes in Liver function markers | Week 0 and week 6
  Alanine transaminase (ALAT) (U/L), Aspartate transaminase (ASAT) (U/L)
Changes in circulating endotoxin/lipopolysaccharide (LPS) concentrations | Week 0 and Week 6
  LPS (pg/ml)
Changes in gut microbiota composition | Week 0 and Week 6
  Measured on fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Mads V Lind, PhD, Principal Investigator — University of Copenhagen, Department of Nutrition, Exercise and Sports
Locations (1):
- University of Copenhagen, Frederiksberg, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No